CLINICAL TRIAL: NCT05836259
Title: First-in-Human, Open-Label, Safety, Tolerability, Dose-Finding, Pharmacodynamic and Cardiac Transgene Expression Study of TN-201, a Recombinant Adeno-associated Virus Serotype 9 (AAV9) Containing Myosin Binding Protein C Transgene, in Adults With MYBPC3 Mutation-associated Hypertrophic Cardiomyopathy (HCM)
Brief Title: Multi-center, Open-label, Single-ascending Dose Study of Safety and Tolerability of TN-201 in Adults With Symptomatic MYBPC3 Mutation-associated HCM
Acronym: MyPEAK-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tenaya Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TN-201-0009
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy (HCM); Myosin Binding Protein C3 (MYBPC3); Nonobstructive HCM; Genetic HCM; Familial HCM; Adenoassociated Virus (AAV); Gene Therapy; Obstructive HCM; nHCM; oHCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Hypertrophic, Familial

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, non-randomized, open label Phase 1b/2 study. The study will consist of 2 escalating dose cohorts. The study will enroll at least 6 and as many as 30 patients. All patients will receive active drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Dose for Cohort 1 will be 3E13 vg/kg
  Interventions: Genetic: TN-201
- Cohort 2 (Experimental): Dose for Cohort 2 will be 6E13 vg/kg
  Interventions: Genetic: TN-201

INTERVENTIONS:
Genetic: TN-201 — TN-201 is a recombinant adeno-associated virus serotype 9 (AAV9) containing Myosin Binding Protein C (MYBPC3) transgene. It is a single (one-time) intravenous dose.

SUMMARY:
This is a first-in-human, non-randomized, open-label study designed to evaluate the safety, tolerability, and pharmacodynamics (PD) of TN-201 in adult patients with symptomatic hypertrophic cardiomyopathy (HCM) caused by mutations in the MYBPC3 gene.

DETAILED DESCRIPTION:
The study will consist of 2 escalating dose cohorts (groups). The study will enroll at least 6 and as many as 30 patients. All patients will receive active drug (TN-201 Gene Therapy). The study will follow patients for 5 years following a single dose of TN-201.

ELIGIBILITY:
Inclusion Criteria:

* MYBPC3 mutation
* Hypertrophic Cardiomyopathy (obstructive and nonobstructive)
* Left Ventricular Ejection Fraction ≥45%
* NYHA Functional Class II or III symptoms
* NT-proBNP ≥160pg/ml

Exclusion Criteria:

* High AAV9 neutralizing antibody titer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Number and severity of Adverse Events over the course of the study. | 5 Years
Number of Serious Adverse Events related to study drug. | 5 Years

SECONDARY OUTCOMES:
Change from baseline to Week 52 in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS). | 52 Weeks
  The score ranges from 0-100, with zero being a worse outcome

OTHER OUTCOMES:
Expression levels of vector genomes and transgene messenger ribonucleic acid (mRNA) and MyBP-C protein in right ventricular (RV) septal biopsy samples at Pre-Treatment, Week 26, and Week 52. | 52 Weeks
Change from Pre-Treatment period in N-terminal pro B-type natriuretic peptide (NTproBNP), and high-sensitivity cardiac troponin I (hs-cTnI) levels. | 5 Years
Percentage of patients who had a change in New York Heart Association (NYHA) Functional Class from baseline. | 5 Years
Change from baseline in echocardiography measurements of indexed left atrial and left ventricular (LV) volumes. | 5 Years
Change from baseline in echocardiography measurements of LV mass. | 5 Years
Change from baseline in echocardiography measurements of maximal LV wall thickness. | 5 Years
Change from baseline in echocardiography measurements of global longitudinal strain. | 5 Years
Change from baseline in 6MWT distance. | 5 Years
Change from baseline peak exercise capacity (pVO2). | 5 Years

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UC San Diego Altman Clinical and Translational Research Institute - Center for Clinical Research, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Christ Hospital Physicians - The Ohio Heart and Vascular Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Grisorio L, Bongianino R, Gianeselli M, Priori SG. Gene therapy for cardiac diseases: methods, challenges, and future directions. Cardiovasc Res. 2024 Nov 25;120(14):1664-1682. doi: 10.1093/cvr/cvae207. PMID 39302117